CLINICAL TRIAL: NCT03851484
Title: Sensory Symptoms in Tourette Syndrome
Acronym: SenST
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Isaacs, Associate Professor of Neurology, Vanderbilt University Medical Center
Other Study IDs: VUMCSenST
Record Dates: First submitted 2019-02-17; First posted 2019-02-22 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Tourette Syndrome
Keywords: Tourette syndrome; premonitory urge; sensory dysregulation; hypersensitivity
MeSH Terms: conditions — Tourette Syndrome; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patients with tics will be asked to complete a series of validated questionnaires (in electronic and/or paper format) regarding symptoms and conditions often associated with Tourette syndrome, including premonitory urges, sensory experiences, inattention, obsessive-compulsive tendencies, anxiety, and depression. Participants will also be asked to complete a quality of life assessment. This series of questionnaires will be administered annually.

DETAILED DESCRIPTION:
Patients with tics will be recruited to participate in an observational study assessing extent and variation in non-motor features of Tourette syndrome over time. Each participant will complete a battery of validated questionnaires and scales online or in paper format (per patient preference), including the Premonitory Urge to Tic Scale (PUTS), the Sensory Gating Inventory (SGI), the Sensory Perception Quotient, the ADHD Self-Report Screening Scale, and others. These questionnaires will be administered annually to patients. For the analysis, participants will be stratified by age into late adolescents (18-25 years old) and adults (older than 25 years) since adolescent development ends at approximately age 25.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older
* Ability to provide informed consent and answer self-report questionnaires independently in English
* Diagnosis of Tourette syndrome (TS), chronic motor tic disorder, or chronic vocal tic disorder

Exclusion criteria:

* History of psychotic disorder
* History of significant neurologic disorder (e.g., stroke) other than TS or another chronic tic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals 18 years and older with Tourette syndrome or other chronic tic disorder
Sampling Method: Non-Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline Sensory Perception Quotient score, short form | Initial assessment at enrollment (time zero)
  Validated instrument assessing anomalous sensory experiences. Scale consists of 35 items screening patients for hyper- or hypo-sensitivity to each of the sensory domains (touch, sight, sound, smell, and taste). Each scale item is a statement to which participants provide a ranking:
  0 = strongly agree
  1. = agree
  2. = disagree
  3. = strongly disagree The minimum score on the short from is 0; the maximum score is 140. Higher scores indicate more abnormal sensory experiences.
Change in Sensory Perception Quotient score, short form at 1 year | 1 year
  Validated instrument assessing anomalous sensory experiences. Scale consists of 35 items screening patients for hyper- or hypo-sensitivity to each of the sensory domains (touch, sight, sound, smell, and taste). Each scale item is a statement to which participants provide a ranking:
  0 = strongly agree
  1. = agree
  2. = disagree
  3. = strongly disagree The minimum score on the short from is 0; the maximum score is 140. Higher scores indicate more abnormal sensory experiences.
Change in Sensory Perception Quotient score, short form at 2 years | 2 years
  Validated instrument assessing anomalous sensory experiences. Scale consists of 35 items screening patients for hyper- or hypo-sensitivity to each of the sensory domains (touch, sight, sound, smell, and taste). Each scale item is a statement to which participants provide a ranking:
  0 = strongly agree
  1. = agree
  2. = disagree
  3. = strongly disagree The minimum score on the short from is 0; the maximum score is 140. Higher scores indicate more abnormal sensory experiences.

SECONDARY OUTCOMES:
Change in Sensory Gating Inventory score at 2 years | 2 years
  Validated instrument assessing anomalous sensory experiences. The scale consists of 36 items screening patients for hyper- or hypo-sensitivity to several of the sensory domains (primarily sight and sound). Each scale item is a statement to which participants provide a ranking:
  1. = never true
  2. = infrequently true
  3. = sometimes but infrequently true
  4. = sometimes true
  5. = true
  6. = always true The minimum score on the scale is 36; the maximum score is 216. Higher scores indicate more abnormal sensory experiences.
Change in Sensory Gating Inventory score at 1 year | 1 year
  Validated instrument assessing anomalous sensory experiences. The scale consists of 36 items screening patients for hyper- or hypo-sensitivity to several of the sensory domains (primarily sight and sound). Each scale item is a statement to which participants provide a ranking:
  1. = never true
  2. = infrequently true
  3. = sometimes but infrequently true
  4. = sometimes true
  5. = true
  6. = always true The minimum score on the scale is 36; the maximum score is 216. Higher scores indicate more abnormal sensory experiences.
Baseline Sensory Gating Inventory score | Initial assessment at enrollment (time zero)
  Validated instrument assessing anomalous sensory experiences. The scale consists of 36 items screening patients for hyper- or hypo-sensitivity to several of the sensory domains (primarily sight and sound). Each scale item is a statement to which participants provide a ranking:
  1. = never true
  2. = infrequently true
  3. = sometimes but infrequently true
  4. = sometimes true
  5. = true
  6. = always true The minimum score on the scale is 36; the maximum score is 216. Higher scores indicate more abnormal sensory experiences.
Change in Premonitory Urge to Tic Scale score at 2 years | 2 years
  Validated instrument assessing type and extent of premonitory sensations. The scale consists of 9 scored items and 1 non-scored item, all assessing degree of abnormal sensations and urges preceding a tic. The scored scale items are ranked 1-4, with 4 being the most abnormal. The minimum score on the scale is 9; the maximum score is 36. Higher scores indicate more frequent and severe premonitory urges.
Change in Premonitory Urge to Tic Scale score at 1 year | 1 year
  Validated instrument assessing type and extent of premonitory sensations. The scale consists of 9 scored items and 1 non-scored item, all assessing degree of abnormal sensations and urges preceding a tic. The scored scale items are ranked 1-4, with 4 being the most abnormal. The minimum score on the scale is 9; the maximum score is 36. Higher scores indicate more frequent and severe premonitory urges.
Baseline Premonitory Urge to Tic Scale score | Initial assessment at enrollment (time zero)
  Validated instrument assessing type and extent of premonitory sensations. The scale consists of 9 scored items and 1 non-scored item, all assessing degree of abnormal sensations and urges preceding a tic. The scored scale items are ranked 1-4, with 4 being the most abnormal. The minimum score on the scale is 9; the maximum score is 36. Higher scores indicate more frequent and severe premonitory urges.

OTHER OUTCOMES:
Yale Global Tic Severity Scale Total Tic Score at baseline | Initial assessment at enrollment (time zero)
  Validated, gold-standard clinician-administered tic assessment scale, comprised of 11 items. Scale range: 0 (best) - 100 (worst)
Change in Yale Global Tic Severity Scale Total Tic Score at 1 year | 1 year
  Validated, gold-standard clinician-administered tic assessment scale, comprised of 11 items. Scale range: 0 (best) - 100 (worst)
Change in Yale Global Tic Severity Scale Total Tic Score at 2 years | 2 years
  Validated, gold-standard clinician-administered tic assessment scale, comprised of 11 items. Scale range: 0 (best) - 100 (worst)
Dimensional Obsessive Compulsive Scale (DOCS) at baseline | Initial assessment at enrollment (time zero)
  Validated self-report questionnaire assessing severity of obsessive and compulsive symptoms, comprised of 20 items. Scale range 0 (least affected) - 80 (most affected)
Dimensional Obsessive Compulsive Scale (DOCS) at 1 year | 1 year
  Validated self-report questionnaire assessing severity of obsessive and compulsive symptoms, comprised of 20 items. Scale range 0 (least affected) - 80 (most affected)
Dimensional Obsessive Compulsive Scale (DOCS) at 2 years | 2 years
  Validated self-report questionnaire assessing severity of obsessive and compulsive symptoms, comprised of 20 items. Scale range 0 (least affected) - 80 (most affected)
Adult ADHD Self-Report Screening Scale for DSM-5 at baseline | Initial assessment at enrollment (time zero)
  Validated self-report scale, developed since release of Diagnostic and Statistical Manual-V, comprised of 6 items. Scale range 0 (least affected) - 24 (most affected)
Adult ADHD Self-Report Screening Scale for DSM-5 at 1 year | 1 year
  Validated self-report scale, developed since release of Diagnostic and Statistical Manual-V, comprised of 6 items. Scale range 0 (least affected) - 24 (most affected)
Adult ADHD Self-Report Screening Scale for DSM-5 at 2 years | 2 years
  Validated self-report scale, developed since release of Diagnostic and Statistical Manual-V, comprised of 6 items. Scale range 0 (least affected) - 24 (most affected)
Gilles de la Tourette Syndrome - Quality of Life Scale (GTS-QOL) at baseline | Initial assessment at enrollment (time zero)
  Validated self-report questionnaire assessing health-related quality of life for patients with Tourette syndrome, comprised of 27 items. Scale range 0 (best quality of life) - 108 (worst quality of life)
Gilles de la Tourette Syndrome - Quality of Life Scale (GTS-QOL) at 1 year | 1 year
  Validated self-report questionnaire assessing health-related quality of life for patients with Tourette syndrome, comprised of 27 items. Scale range 0 (best quality of life) - 108 (worst quality of life)
Gilles de la Tourette Syndrome - Quality of Life Scale (GTS-QOL) at 2 years | 2 years
  Validated self-report questionnaire assessing health-related quality of life for patients with Tourette syndrome, comprised of 27 items. Scale range 0 (best quality of life) - 108 (worst quality of life)
Multidimensional Assessment of Interoceptive Awareness-2 (MAIA-2) at baseline | Initial assessment at enrollment (time zero)
  Validated self-report questionnaire assessing interoceptive sensibility, comprised of 37 items. Each scale item is a statement to which respondents must select "never" (0) to "always" (5) on a six-point Likert scale. No total MAIA-2 score exists. Rather, individual scale items belong to one of eight MAIA-2 subscales. For each subscale, higher score signifies more of that construct.
Multidimensional Assessment of Interoceptive Awareness-2 (MAIA-2) at 1 year | 1 year
  Validated self-report questionnaire assessing interoceptive sensibility, comprised of 37 items. Each scale item is a statement to which respondents must select "never" (0) to "always" (5) on a six-point Likert scale. No total MAIA-2 score exists. Rather, individual scale items belong to one of eight MAIA-2 subscales. For each subscale, higher score signifies more of that construct.
Multidimensional Assessment of Interoceptive Awareness-2 (MAIA-2) at 2 years | 2 years
  Validated self-report questionnaire assessing interoceptive sensibility, comprised of 37 items. Each scale item is a statement to which respondents must select "never" (0) to "always" (5) on a six-point Likert scale. No total MAIA-2 score exists. Rather, individual scale items belong to one of eight MAIA-2 subscales. For each subscale, higher score signifies more of that construct.
Body Perception Questionnaire - Short Form (BPQ-SF) at baseline | Initial assessment at enrollment (time zero)
  Validated self-report questionnaire assessing interoceptive sensibility, comprised of 46 items total, divided into 3 sections: Body Awareness (raw total score 26-130), Supradiaphragmatic Reactivity (raw total score 15-69), and Subdiaphragmatic Reactivity (raw total score 6-28). Raw scores are converted to T-scores. Higher raw and T-scores indicate greater maladaptive body awareness.
Body Perception Questionnaire - Short Form (BPQ-SF) at 1 year | 1 year
  Validated self-report questionnaire assessing interoceptive sensibility, comprised of 46 items total, divided into 3 sections: Body Awareness (raw total score 26-130), Supradiaphragmatic Reactivity (raw total score 15-69), and Subdiaphragmatic Reactivity (raw total score 6-28). Raw scores are converted to T-scores. Higher raw and T-scores indicate greater maladaptive body awareness.
Body Perception Questionnaire - Short Form (BPQ-SF) at 2 years | 2 year
  Validated self-report questionnaire assessing interoceptive sensibility, comprised of 46 items total, divided into 3 sections: Body Awareness (raw total score 26-130), Supradiaphragmatic Reactivity (raw total score 15-69), and Subdiaphragmatic Reactivity (raw total score 6-28). Raw scores are converted to T-scores. Higher raw and T-scores indicate greater maladaptive body awareness.
Generalized Anxiety Disorder 7 (GAD-7) at baseline | Initial assessment at enrollment (time zero)
  Validated self-report scale for anxiety, comprised of 7 items. Scale range 0 (least severe) - 21 (most severe).
Generalized Anxiety Disorder 7 (GAD-7) at 1 year | 1 year
  Validated self-report scale for anxiety, comprised of 7 items. Scale range 0 (least severe) - 21 (most severe).
Generalized Anxiety Disorder 7 (GAD-7) at 2 years | 2 years
  Validated self-report scale for anxiety, comprised of 7 items. Scale range 0 (least severe) - 21 (most severe).
Patient Health Questionnaire 9 (PHQ-9) at baseline | Initial assessment at enrollment (time zero)
  Validated self-report scale for depression, comprised of 9 items. Scale range 0 (least severe) - 27 (most severe).
Patient Health Questionnaire 9 (PHQ-9) at 1 year | 1 year
  Validated self-report scale for depression, comprised of 9 items. Scale range 0 (least severe) - 27 (most severe).
Patient Health Questionnaire 9 (PHQ-9) at 2 years | 2 years
  Validated self-report scale for depression, comprised of 9 items. Scale range 0 (least severe) - 27 (most severe).

CONTACTS AND LOCATIONS:
Overall Officials: David A Isaacs, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Isaacs D, Key AP, Cascio CJ, Conley AC, Riordan H, Walker HC, Wallace MT, Claassen DO. Cross-disorder comparison of sensory over-responsivity in chronic tic disorders and obsessive-compulsive disorder. Compr Psychiatry. 2022 Feb;113:152291. doi: 10.1016/j.comppsych.2021.152291. Epub 2021 Dec 17. PMID 34952304
- [Background] Isaacs DA, Riordan HR, Claassen DO. Clinical Correlates of Health-Related Quality of Life in Adults With Chronic Tic Disorder. Front Psychiatry. 2021 Mar 10;12:619854. doi: 10.3389/fpsyt.2021.619854. eCollection 2021. PMID 33776814
- [Background] Isaacs D, Key AP, Cascio CJ, Conley AC, Walker HC, Wallace MT, Claassen DO. Sensory Hypersensitivity Severity and Association with Obsessive-Compulsive Symptoms in Adults with Tic Disorder. Neuropsychiatr Dis Treat. 2020 Nov 2;16:2591-2601. doi: 10.2147/NDT.S274165. eCollection 2020. PMID 33173296